CLINICAL TRIAL: NCT01448837
Title: 24-Hour Intraocular Pressure Control Obtained With the Bimatoprost/Timolol Fixed Combination Compared With Latanoprost as First Choice Therapy in Subjects With Exfoliation Syndrome, or Exfoliative Glaucoma
Brief Title: 24-Hour Intraocular Pressure Control With Bimatoprost/Timolol Versus Latanoprost as First Choice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A5134
Record Dates: First submitted 2011-09-26; First posted 2011-10-07 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Bimatoprost; Timolol; Ganfort; Latanoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bimatoprost/Timolol drops (Active Comparator): The patients will be treated with bimatoprost/timolol fixed combination therapy
  Interventions: Drug: Bimatoprost/Timolol, 24-hour intraocular pressure monitoring; Drug: Latanoprost, 24-hour intraocular pressure monitoring
- Latanoprost drops (Active Comparator): The patients will be crossed over to therapy with latanoprost
  Interventions: Drug: Bimatoprost/Timolol, 24-hour intraocular pressure monitoring; Drug: Latanoprost, 24-hour intraocular pressure monitoring

INTERVENTIONS:
Drug: Bimatoprost/Timolol, 24-hour intraocular pressure monitoring — Administered once in the evening
  Other Names: Ganfort; Xalatan
Drug: Latanoprost, 24-hour intraocular pressure monitoring — assessment of 24-hour efficacy for the two drugs after 3 months of chronic dosing
  Other Names: Ganfort; Xalatan

SUMMARY:
The primary objective of this crossover 24-hour Intraocular Pressure (IOP) trial is to compare the control obtained after 3 months of therapy with the bimatoprost/timolol fixed combination (BTFC, Ganfort) given once in the evening (20:00) versus latanoprost (Xalatan) administered once in the evening (20:00) in newly-diagnosed patients with exfoliation syndrome (XFS) and ocular hypertension, or exfoliative glaucoma (XFG) previously untreated and IOP greater than 29 mm Hg.

ELIGIBILITY:
Inclusion Criteria:

* Patient has exfoliation syndrome with ocular hypertension, or exfoliative glaucoma and is older than 29 years
* Patient is newly diagnosed, or currently untreated and exhibits untreated morning IOP (2 separate IOP readings at 10:00)greater than 29 mm Hg in the study eye
* Study patients should have mild to moderate exfoliative glaucoma (VF loss <12 dB; cupping 0.8 or less)
* Patient with exfoliation syndrome should fulfill the IOP criterion (IOP > 29 mm Hg at 10:00)
* Patient deemed by investigator to require significant IOP reduction to obtain desired target IOP
* Patient agrees to be treated for at least 3 months with latanoprost and bimatoprost/timolol fixed combination drops dosed in the evening
* In study eye distance best corrected Snelen visual acuity greater than 1/10

Exclusion Criteria:

* Contraindications to therapy with latanoprost, bimatoprost, or β-blockers
* History of non-adherence or previously recorded evidence of lack of response (<10% morning IOP reduction) to any antiglaucoma medication
* Patient can not understand the instructions and adhere to medications
* Patient is a female of childbearing potential or lactating mother
* Past history of trauma, inflammation, surgery, past use of steroids (within 2 months), severe dry eyes and use of contact lenses
* Signs of ocular infection, except blepharitis, or corneal abnormality that may affect IOP measurements
* The other eye can not receive the same therapy, or remain without medical therapy
* Closed angles

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
24-hour IOP reduction between the two medications | 3 months
  Bimatoprost/Timolol will obtain a statistically greater 24-hour IOP reduction than latanoprost and the mean 24-hour IOP difference between the two medications will be clinically meaningful (at least 2 mm Hg).

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios G Konstas, MD, PhD, Principal Investigator — Glaucoma Unit, 1st University Department of Ophthalmology
Locations (1):
- Glaucoma Unit, 1st University Department of Ophthalmology, Thessaloniki, Greece